CLINICAL TRIAL: NCT01891643
Title: A Phase 3, Randomized, Open Label Trial of Lenalidomide/Dexamethasone With or Without Elotuzumab in Subjects With Previously Untreated Multiple Myeloma
Brief Title: PH III Study of Lenalidomide and Dexamethasone With or Without Elotuzumab to Treat Previously Untreated Multiple Myeloma (ELO 1 Substudy)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CA204-006 (Biomarker Substudy); 2010-022445-20 (EudraCT Number)
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Results first posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Newly Diagnosed, Previously Untreated Multiple Myeloma
MeSH Terms: interventions — Lenalidomide; Dexamethasone; Calcium Dobesilate; elotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Lenalidomide + Dexamethasone (Experimental): Lenalidomide 25 mg capsules by mouth once daily (on Days 1-21), repeat every 28 days until subject meets criteria for discontinuation of study drug
  Dexamethasone 40 mg tablets by mouth weekly (on Days 1, 8, 15, 22), repeat every 28 days until subject meets criteria for discontinuation of study drug
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone
- Arm 2: Lenalidomide + Dexamethasone + Elotuzumab (Experimental): Lenalidomide 25 mg capsules by mouth once daily (Days 1-21)
  Dexamethasone 28 mg tablets by mouth once daily [Days 1, 8, 15, 22 (cycles 1 & 2); Days 1 & 15(cycles 3-18); Day 1 (cycle 19 & beyond)]
  Dexamethasone 40 mg tablets by mouth once daily [Days 8 & 22 (cycles 3-18); Days 8, 15, 22 (cycle 19 & beyond)]
  Dexamethasone 8 mg IV (intravenous) solution once daily [Days 1, 8, 15, 22 (cycles 1 & 2); Days 1 & 15 (cycles 3-18); Day 1 (cycle 19 & beyond)]
  Elotuzumab 10 mg/kg IV solution weekly [Days 1, 8, 15, 22 (cycles 1 & 2); Days 1 & 15 (cycles 3-18)]
  Elotuzumab 20 mg/kg IV solution on Day 1 (cycle 19 & beyond)
  Repeat above-mentioned dose cycles every 28 days until subject meets criteria for discontinuation of study drug
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Biological: Elotuzumab

INTERVENTIONS:
Drug: Lenalidomide
  Other Names: Revlimid®
Drug: Dexamethasone
  Other Names: Decadron®; Dexamethasone Intensol®; Dexpak®; Taperpak®
Biological: Elotuzumab
  Other Names: BMS-901608
  Arms: Arm 2: Lenalidomide + Dexamethasone + Elotuzumab

SUMMARY:
The purpose of the study is to look at subjects who receive Lenalidomide, Dexamethasone, and Elotuzumab and determine if they will have lower surface CS1 expression on malignant plasma cells at the time of progression than those who receive Lenalidomide and Dexamethasone without Elotuzumab

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

Subjects who are newly diagnosed with symptomatic MM and who:

* Have not received any prior systemic anti-myeloma therapy
* Have measurable disease
* And are not candidates for high-dose therapy plus stem-cell transplantation (SCT) because of age (≥65 years) or coexisting conditions. Refusal to undergo high dose therapy with SCT is NOT sufficient for entry onto CA204-006 for a subject <65 years old. There must be a comorbidity that prevents SCT for a subject <65 years old

Exclusion Criteria:

* Subjects with non-secretory or oligo-secretory or free light-chain only myeloma
* Smoldering MM, defined as asymptomatic MM with absence of lytic bone lesions
* Monoclonal Gammopathy of Undetermined Significance (MGUS)
* Active plasma cell leukemia
* Known Human Immunodeficiency Virus (HIV) infection or active hepatitis A, B, or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- United States (9):
  - Pacific Hematology Oncology Associates, San Francisco, California
  - Memorial Cancer Institute, Hollywood, Florida
  - Illinois Cancercare, Pc, Peoria, Illinois
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - Crescent City Research Consortium, LLC, Marrero, Louisiana
  - Ohio State University Medical Center, Columbus, Ohio
  - Medical University Of South Carolina Hollings Cancer Center, Charleston, South Carolina
  - Baptist Cancer Center, Memphis, Tennessee
  - Northern Utah Associates, Ogden, Utah
- Local Institution, Athens, Greece
- Italy (2):
  - Local Institution, Genova
  - Local Institution, Rome
- Poland (2):
  - Local Institution, Chorzów
  - Local Institution, Lublin

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 23 participants treated in the main CA204-006 study (NCT01335399) were recruited for the CA204-006 biomarker sub-study (NCT01891643).
  No additional treatment (other than what administered in the main study) was dosed during the biomarker sub-study.
Groups:
- E-Ld Cohort: Participants receiving a combination of Elotuzumab (E) Lenalidomide (L) Dexamethasone (d) in a 28 day cycle
- Ld Cohort: Participants receiving a combination of Lenalidomide (L) Dexamethasone (d) in a 28 day cycle
Period: Overall Study
Arm/Group | E-Ld Cohort | Ld Cohort
Started | 13 | 10
Completed (Completed = continuing treatment in the main CA204-006 study (NCT01335399)) | 3 | 0
Not Completed | 10 | 10
Not completed — Adverse event unrelated to study drug | 2 | 5
Not completed — Disease Progression | 4 | 3
Not completed — Study Drug Toxicity | 3 | 0
Not completed — Maximum Clinical Benefit | 0 | 1
Not completed — Poor/Non-compliance | 0 | 1
Not completed — Participant request to discontinue | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E-Ld Cohort | Ld Cohort | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.8 (6.77) | 71.3 (6.53) | 73.3 (6.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 11 | 7 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 12 | 9 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Progression of the Cell Surface Expression of CS1 From Bone Marrow-Derived Multiple Myeloma (MM) Cells
Description: CS1 (CD2 subset-1, also known as CRACC, SLAMF7, CD319) expression levels in multiple myeloma cells were analyzed from bone-marrow aspirates collected at baseline and at time of progression through mean fluorescent intensity.
  The following conditions were considered to describe multiple myeloma cells expressing CS1 (CS1+/CD38++/CD138+/CD56+/CD19-/CD45DIM)
Time Frame: From baseline (screening) to time of progression (up to approximately 54 months)
Population: All treated participants with measurements available at baseline and at time of progression.
  No participants in any of the 2 cohorts had available measurements both at baseline and time of progression
Arm/Group | E-Ld Cohort | Ld Cohort
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percent of Bone Marrow-Derived Multiple Myeloma (MM) Cells Expressing Cell Surface CS1 at Time of Progression
Description: CS1 (CD2 subset-1, also known as CRACC, SLAMF7, CD319) expression levels in multiple myeloma cells were analyzed from bone-marrow aspirates collected at time of progression.
  The following conditions were considered to describe multiple myeloma cells expressing CS1 (CS1+/CD38++/CD138+/CD56+/CD19-/CD45DIM)
Time Frame: Time of progression (up to approximately 54 months from pre-treatment screening)
Population: All treated participants with measurements available at time of progression.
Measure: Median (Full Range); unit: Percent of cells expressing CS1
Arm/Group | E-Ld Cohort | Ld Cohort
Number analyzed (Participants) | 4 | 1
Percent of cells expressing CS1 | 46.59 [0.0 to 99.1] | 84.62 [NA to NA] — Only 1 participant analyzed

3. Secondary Outcome: Levels of CS1 Soluble Form (sCS1) in Serum
Description: Expression levels of the free form of soluble CS1 were analyzed at different timepoints from serum samples derived from peripheral blood collection
Time Frame: At baseline (screening), during main study therapy (cycle 3 day 1, up to 64 days) and at time of progression (up to approximately 31 months)
Population: All treated participants with measurements available either at baseline, at cycle 3 day 1 of study therapy or at time of progression.
Measure: Median (Full Range); unit: ug/L
Arm/Group | E-Ld Cohort | Ld Cohort
Number analyzed (Participants) | 13 | 10
ug/L
  Baseline: number analyzed (Participants) | 11 | 7
  Baseline | 3.60 [0.7 to 7.4] | 13.27 [2.2 to 79.8]
  Cycle 3 day 1 of main study therapy: number analyzed (Participants) | 7 | 4
  Cycle 3 day 1 of main study therapy | 0.15 [0.1 to 0.3] | 0.72 [0.2 to 3.0]
  Time of progression: number analyzed (Participants) | 3 | 1
  Time of progression | 0.39 [0.2 to 0.5] | 49.85 [NA to NA] — Only 1 participant analyzed

4. Secondary Outcome: Change From Baseline in the Levels of CS1 Soluble Form (sCS1) in Serum During Therapy and At Progression
Description: as for outcome 3
Time Frame: From baseline (screening) to cycle 3 day 1 of the main study therapy (up to 64 days) and from baseline (screening) to time of progression (up to approximately 31 months)
Population: All treated participants with measurements available at baseline and at cycle 3 day 1 of study therapy or at baseline and at the time of progression.
Measure: Median (Full Range); unit: ug/L
Arm/Group | E-Ld Cohort | Ld Cohort
Number analyzed (Participants) | 13 | 10
ug/L
  From baseline to Cycle 3 day 1 of main study therapy: number analyzed (Participants) | 7 | 4
  From baseline to Cycle 3 day 1 of main study therapy | -3.51 [-6.9 to -0.6] | -4.08 [-15.1 to -1.6]
  From baseline to time of progression: number analyzed (Participants) | 3 | 1
  From baseline to time of progression | -0.85 [-6.9 to -0.4] | -17.41 [NA to NA] — Only 1 participant analyzed

5. Secondary Outcome: Change From Baseline in the Number of Circulating Multiple Myeloma (MM) Cells
Description: Circulating MM cells isolated from peripheral blood
Time Frame: From baseline (screening) to cycle 3 day 1 of the main study therapy (up to 64 days) and from baseline (screening) to the time of progression (up to approximately 54 months)
Population: All treated participants with available circulating MM cells. Circulating MM cells were not collected for any of the participants.
Arm/Group | E-Ld Cohort | Ld Cohort
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Cell Surface CS1 Expression Levels in Circulating Multiple Myeloma (MM) Cells
Description: Circulating MM cells isolated from peripheral blood
Time Frame: as for outcome 5
Population: All treated participants with available circulating MM cells and CS1 expression levels.
  Circulating MM cells were not collected for any of the participants.
Arm/Group | E-Ld Cohort | Ld Cohort
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: CS1 Expression Levels in Matched Samples of Bone Marrow-Derived Multiple Myeloma (MM) Cells and Circulating MM Cells
Description: CS1 expression levels analyzed from matching bone marrow aspirates (for bone marrow-derived MM cells) and from peripheral blood (for circulating tumor cells) collected from the same participants
Time Frame: At baseline (screening), during main study therapy (cycle 3 day 1) and at time of progression (up to approximately 54 months)
Population: All treated participants with matched samples of bone marrow-derived MM cells and circulating MM cells.
  Circulating MM cells were not collected for any of the participants.
Arm/Group | E-Ld Cohort | Ld Cohort
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose to 60 days following last dose (up to approximately 80 months)
Arm/Group | E-Ld Cohort | Ld Cohort
All-Cause Mortality (participants affected / at risk) | 8/13 | 5/10
Serious Adverse Events (participants affected / at risk) | 9/13 | 7/10
Other Adverse Events (participants affected / at risk) | 13/13 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E-Ld Cohort (N=13) | Ld Cohort (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Refractory anaemia with ringed sideroblasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Delusional disorder, unspecified type (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E-Ld Cohort (N=13) | Ld Cohort (N=10)
Anaemia (Blood and lymphatic system disorders) | 3 | 6
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 2 | 1
Macular degeneration (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3
Retching (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 0 | 2
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 6 | 2
Fibrosis (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 5
Pyrexia (General disorders) | 1 | 3
Hypersensitivity (Immune system disorders) | 2 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 2
Conjunctivitis (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1
Genitourinary tract infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 2
Intervertebral discitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Onychomycosis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 2 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood albumin decreased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 2 | 1
Blood lactate dehydrogenase decreased (Investigations) | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 0 | 1
Creatinine renal clearance decreased (Investigations) | 1 | 0
Glomerular filtration rate decreased (Investigations) | 2 | 2
Neutrophil count decreased (Investigations) | 1 | 2
Neutrophil count increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 2 | 0
Weight increased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Carotid arteriosclerosis (Nervous system disorders) | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1
Sciatica (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Spinal cord herniation (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 1 | 2
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 3
Mood altered (Psychiatric disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Glomerulonephritis minimal lesion (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2013-02-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT01891643/Prot_000.pdf
  • Statistical Analysis Plan (2013-02-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT01891643/SAP_001.pdf